CLINICAL TRIAL: NCT05329389
Title: Adherence to Fluid Intake Recommendations After Stone Removal in Low Risk Group Patients
Brief Title: Adherence to Fluid Intake Recommendations in Kidney Stone Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gadzhiev Nariman (Other)
Responsible Party: Sponsor-Investigator, Gadzhiev Nariman, PhD, Urologist, Deputy Medical Director of Saint-Petersburg State University Clinic, Saint Petersburg State University, Russia
Organization: Saint Petersburg State University, Russia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: StoneMD_Schools_for_patients
Record Dates: First submitted 2022-03-29; First posted 2022-04-15 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Urolithiasis
Keywords: application; StoneMD; Schools of patients
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: In case of presence/absence of inclusion/exclusion criteria and written informed consent will be obtained, patients will be randomized in a 1:1:1 ratio according to the list of randomized blocks using a computer generator. Patients will be randomized at the last available moment in order to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- StoneMD (Experimental): Patients will receive standard recommendations of keeping diuresis at the level of 2.5 l/day and to use the StoneMD application on their smartphones after the surgery. Patients will use the section "Water balance" and follow the instructions during the 12 month after the surgery.
  Interventions: Device: StoneMD; Behavioral: Standard recommendation
- StoneMD & Schools of Patients (Experimental): Patients will receive standard recommendations of keeping diuresis at the level of 2.5 l/day and and recommendations to use the StoneMD application on their smartphones after the surgery. Patients will use the section "Water balance" and follow the instructions during the 12 month after the surgery. Additionally, patients will visit schools during a following year. Patients receive 4 consultations (one per 3 month).
  Interventions: Device: StoneMD; Behavioral: Schools of Patients; Behavioral: Standard recommendation
- Recommendations only (Active Comparator): Only fluid balance recommendations given at the day of discharge. Patients will receive recommendations of keeping diuresis at the level of 2.5 l/day after the surgery
  Interventions: Behavioral: Standard recommendation

INTERVENTIONS:
Device: StoneMD — StoneMD - is an app from App Store (for iOS) or Google Play (for Android).
  Arms: StoneMD; StoneMD & Schools of Patients
Behavioral: Schools of Patients — The "Schools for Patients" with Urolithiasis is an online course for patients with urinary stone disease.
  Arms: StoneMD & Schools of Patients
Behavioral: Standard recommendation — Only fluid balance recommendations given at the day of discharge.

SUMMARY:
The cumulative risk of stone recurrence rate is up to 14% at 1 year, 35% at 5 years, and 52% at 10 years. Low urine volume caused by insufficient fluid consumption is one of the most crucial risk factors for kidney stone formation. According to the guidelines, a copious fluid intake to maintain a urine volume of at least 2.0 to 2.5 L/24 h is recommended for most kidney stone formers. Patients often find it difficult to follow the recommendations in fluid intake, which leads to stone recurrence. Therefore, there is a need to improve patient compliance and adherence to following the instructions on keeping water balance. For this purpose we developed a mixed educational program including two parts. The first is the mobile application called "StoneMD: Kidney Stones". The second is the "School for Patients" with kidney stones, which is responsible for the stone clinic effect.

DETAILED DESCRIPTION:
The aim of the study is to test the hypothesis that using mixed educational program additionally to standard recommendations in patients after the first stone surgery episode helps to achieve better adherence to daily fluid intake recommendations than the using standard recommendations alone given at the day of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Low risk recurrence group patients;
* Patients after the first stone surgery;

Exclusion Criteria:

* Recurrent cases of stone formation;
* Patients, who do not have smartphones;
* Patients, who can't visit "Schools for Patients" with kidney stone disease;

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-04 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Volume of daily urine | 12 month after the surgery
  The primary outcome will be measured in the lab in international units of measurement
Concentration of creatinine in daily urine | 12 month after the surgery
  The primary outcome will be measured in the lab in international units of measurement

SECONDARY OUTCOMES:
Likert scale questionnaire scores | 12 month
  Likert scale questionnaire of the usefulness of the app "StoneMD" and "Schools for patients". Higher scores means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nariman Gadzhiev, PhD, Principal Investigator — Deputy Medical Director
Locations (1):
- SBPSU, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uribarri J, Oh MS, Carroll HJ. The first kidney stone. Ann Intern Med. 1989 Dec 15;111(12):1006-9. doi: 10.7326/0003-4819-111-12-1006. PMID 2688503
- [Background] Siener R, Hesse A. Fluid intake and epidemiology of urolithiasis. Eur J Clin Nutr. 2003 Dec;57 Suppl 2:S47-51. doi: 10.1038/sj.ejcn.1601901. PMID 14681713
- [Background] Skolarikos A, Straub M, Knoll T, Sarica K, Seitz C, Petrik A, Turk C. Metabolic evaluation and recurrence prevention for urinary stone patients: EAU guidelines. Eur Urol. 2015 Apr;67(4):750-63. doi: 10.1016/j.eururo.2014.10.029. Epub 2014 Nov 20. PMID 25454613
- [Background] Becker B, Gadzhiev N, Popiolek M, Gross AJ, Netsch C. [A mobile app for patients suffering from kidney stones]. Urologe A. 2018 May;57(5):577-582. doi: 10.1007/s00120-018-0652-0. German. PMID 29713752
- [Background] Gadjiev N.K., Gorelov D.S., Akopyan G.N., Gelig V.A., Ivanov A.O., Petrov S.B., Kryukova N.U., Reva S.A., Ponomareva Yu.A., Al-Shukri A.S., Mischenko A.A., Kogai M.A., Vasiliev V.N., Chernysheva D.Yu., Obidnyak V.M., Makar'in V.A., Pisarev A.V., Zakuckij A.N., Kuzmin I.V., Amdiy R.E., Korneyev I.A., Al-Shukri S.H. "Schools for Patients" with Urolithiasis and Prostatic Diseases. Vestnik Urologii. 2020;8(1):110-120. (In Russ.) https://doi.org/10.21886/2308-6424-2020-8-1-110-120